CLINICAL TRIAL: NCT04761055
Title: Detection of Breast Lesions Utilizing iBreast Exam: A Comparison With Clinical Breast Exam
Brief Title: Study of iBreast, a Handheld Device to Detect Breast Abnormalities During Screening Visits for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: UE LifeSciences Inc. (Industry); Earlier.org (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-302
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Breast Screening
Keywords: Breast Abnormalities
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Screening Visits for Breast Cancer (Experimental): Consenting patients will receive their already scheduled standard CBE and mammogram and in addition will receive a breast exam utilizing the iBreast Exam (iBE).
  Interventions: Other: Clinical Breast exam (CBE); Device: iBreastExam device; Diagnostic Test: mammogram

INTERVENTIONS:
Other: Clinical Breast exam (CBE) — The standard CBE will be performed by a nurse practitioner (NP) who will record any positive CBE finding.
Device: iBreastExam device — The iBE is an FDA 510(k) cleared portable device which utilizes an array of dynamic capacitive pressure sensors to perform electronic palpation for breast abnormalities. The iBE exam will be administered by a mammogram technologist, blinded to CBE results.
Diagnostic Test: mammogram — All patients will have routine standard mammographic views performed. Patients with positive iBE and/or CBE findings will have additional mammographic and/or ultrasound imaging to determine if a correlating breast lesion is present using the same standard of care algorithm as is used currently for positive CBE findings.

SUMMARY:
This study will test the iBreastExam device to find out whether it can detect a mass or lump in the breast as accurately as a routine breast cancer screening examination.

The iBreastExam is a handheld device that performs a painless electronic palpation (examination by touch) of the breast. The device is designed to detect breast abnormalities that may require breast imaging and additional clinical examination by a nurse or doctor. The iBreastExam device creates a color map of the breast, with red spots indicating areas that may be abnormal.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Over 18 years of age, able to consent
* RLC patients presenting to RLC or BAIC for mammogram and CBE
* Asymptomatic and symptomatic patients will be included

Exclusion Criteria:

* Male patients
* Patients under 18 years of age, unable to consent
* Pregnant patients
* Lactating patients
* Non-intact skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 309 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Compare the Outcomes of the iBE Examinations to Clinical Breast Examinations (CBE)by Estimating the Sensitivity of the Device Using Imaging Results | approximately one month after imaging scan
  comparing the calculated the sensitivities or the percentage of true positive breast lesions (based on imaging results) of the iBE and CBE
Compare the Outcomes of the iBE Examinations to Clinical Breast Examinations by Estimating the Specificity of the Device Using Imaging Results | approximately one month after imaging scan
  comparing the calculated the specificities or the percentage of true negative lesions (based on imaging results) of the iBE and CBE

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Mango, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - MSK at Ralph Lauren (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm